CLINICAL TRIAL: NCT01261793
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study of the Efficacy and Safety of Four 12-week Treatment Cycles (48 Weeks Total) of Epratuzumab in Systemic Lupus Erythematosus Subjects With Moderate to Severe Disease
Brief Title: Study of Epratuzumab Versus Placebo in Subjects With Moderate to Severe General Systemic Lupus Erythematosus (SLE)
Acronym: EMBODY2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL0010; 2010-018565-26 (EudraCT Number)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Monoclonal antibody; B-Cell immunotherapy; Epratuzumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Weekly infusion) (Placebo Comparator): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
  Interventions: Drug: Placebo
- Epratuzumab 600 mg per week (Experimental): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12 week treatment cycles
  Interventions: Drug: Epratuzumab
- Epratuzumab 1200 mg every other week (Experimental): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
  Interventions: Drug: Placebo; Drug: Epratuzumab

INTERVENTIONS:
Drug: Placebo — Placebo infusions delivered weekly for 4 weeks over four 12-week treatment cycles
  Arms: Epratuzumab 1200 mg every other week; Placebo (Weekly infusion)
Drug: Epratuzumab — 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12- week treatment cycles
  Arms: Epratuzumab 600 mg per week
Drug: Epratuzumab — 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles
  Arms: Epratuzumab 1200 mg every other week

SUMMARY:
The primary objective of the study is to confirm the clinical efficacy of epratuzumab in the treatment of subjects with Systemic Lupus Erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Positive antinuclear antibodies (ANA) at Screening (Visit 1)
* Current clinical diagnosis of Systemic Lupus Erythematosus (SLE) by American College of Rheumatology (ACR) criteria such that at least 4 of the 11 criteria are met
* Active moderate to severe SLE activity as demonstrated by the British Isles Lupus Assessment Group Index (BILAG)
* Active moderate to severe SLE disease as demonstrated by SLE disease activity index (SLEDAI) total score
* On stable SLE treatment regimen, including mandatory corticosteroids and immunosuppressants or antimalarials

Exclusion Criteria:

* Subjects who are breastfeeding, pregnant, or plan to become pregnant
* Subjects with active, severe SLE disease activity which involves the renal system
* Subjects with active, severe, neuropsychiatric SLE, defined as any neuropsychiatric element scoring BILAG level A disease.
* Subjects with the evidence of an immunosuppressive state
* Subjects who, in the opinion of the investigator, are at a particularly high risk of significant infection
* History of malignant cancer, except the following treated cancers: cervical carcinoma in situ, basal cell carcinoma, or dermatological squamous cell carcinoma.
* Subjects receiving any live vaccination within the 8 weeks prior to screening (Visit 1).
* Subjects with history of infections, including but not limited to concurrent acute or chronic viral hepatitis B or C
* Subjects with substance abuse or dependence or other relevant concurrent medical condition
* Subjects with history of thromboembolic events within 1 year of screening Visit.
* Subjects with significant hematologic abnormalities
* Subject has received treatment with other anti- B cell antibodies within 12 months prior to screening (visit 1)
* Subject use of oral anticoagulant (not including) nonsteroidal anti-inflammatory drugs (NSAIDs) within 12 weeks prior to screening (Visit 1)
* Subject has previously participated in this study or has previously received epratuzumab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2010-12; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (133):
- United States (49):
  - 539, Birmingham, Alabama
  - 557, Little Rock, Arkansas
  - 515, Hemet, California
  - 544, Huntington Beach, California
  - 550, La Jolla, California
  - 548, Los Angeles, California
  - 589, San Diego, California
  - 531, San Leandro, California
  - 558, Torrance, California
  - 594, Westlake Village, California
  - 532, Denver, Colorado
  - 511, Bridgeport, Connecticut
  - 514, Brandon, Florida
  - 533, Fort Lauderdale, Florida
  - 518, Plantation, Florida
  - 585, Port Orange, Florida
  - 538, Tampa, Florida
  - 537, Atlanta, Georgia
  - 587, Decatur, Georgia
  - 590, Idaho Falls, Idaho
  - 543, Bowling Green, Kentucky
  - 592, Lexington, Kentucky
  - 576, New Orleans, Louisiana
  - 572, Boston, Massachusetts
  - 554, Ann Arbor, Michigan
  - 513, Lansing, Michigan
  - 599, Lansing, Michigan
  - 575, Florissant, Missouri
  - 549, St Louis, Missouri
  - 596, Nashua, New Hampshire
  - 593, Clifton, New Jersey
  - 568, Freehold, New Jersey
  - 551, Brooklyn, New York
  - 553, Lake Success, New York
  - 545, Manhasset, New York
  - 577, Roslyn, New York
  - 559, Charlotte, North Carolina
  - 547, Tulsa, Oklahoma
  - 561, Wyomissing, Pennsylvania
  - 535, Charleston, South Carolina
  - 598, Myrtle Beach, South Carolina
  - 571, Jackson, Tennessee
  - 574, Amarillo, Texas
  - 570, Austin, Texas
  - 541, Houston, Texas
  - 563, Houston, Texas
  - 562, San Antonio, Texas
  - 552, Chesapeake, Virginia
  - 534, Seattle, Washington
- Brazil (5):
  - 954, Belo Horizonte
  - 956, Campinas
  - 955, Goiânia
  - 950, Juiz de Fora
  - 952, Rio de Janeiro
- Canada (7):
  - 506, St. John's, Newfoundland and Labrador
  - 507, Mississauga, Ontario
  - 508, Rimouski, Quebec
  - 502, Hamilton
  - 500, London
  - 504, Toronto
  - 517, Victoria
- France (5):
  - 613, Caen
  - 618, Limoges
  - 617, Montpellier
  - 614, Paris
  - 616, Toulouse
- Germany (12):
  - 628, Berlin
  - 633, Berlin
  - 625, Cologne
  - 636, Dessau
  - 637, Hamburg
  - 632, Herne
  - 629, Kiel
  - 626, Leipzig
  - 634, Mainz
  - 627, Münster
  - 639, Wiesbaden
  - 631, Zerbst
- Hungary (7):
  - 712, Budapest
  - 716, Budapest
  - 718, Budapest
  - 717, Debrecen
  - 711, Szeged
  - 715, Szeged
  - 713, Zalaegerszeg
- India (2):
  - 852, Ahmedabad
  - 853, Bangalore
- Italy (3):
  - 648, Milan
  - 647, Pisa
  - 646, Roma
- Mexico (4):
  - 978, Cuauhtémoc
  - 976, Mexico City
  - 982, México
  - 981, Torreón
- Poland (11):
  - 743, Bydgoszcz
  - 744, Częstochowa
  - 752, Elblag
  - 745, Katowice
  - 746, Katowice
  - 748, Lublin
  - 750, Lublin
  - 742, Poznan
  - 747, Szczecin
  - 751, Ustroń
  - 749, Warsaw
- Romania (6):
  - 757, Bucharest
  - 758, Bucharest
  - 760, Bucharest
  - 759, Constanța
  - 756, Galati
  - 761, Iași
- Russia (3):
  - 778, Kemerovo
  - 780, Kemerovo
  - 779, Moscow
- South Africa (3):
  - 901, Cape Town
  - 902, Durban
  - 903, Stellenbosch
- Spain (6):
  - 661, Barcelona
  - 660, Getafe
  - 662, Las Palmas de Gran Canaria
  - 664, Madrid
  - 663, Santiago de Compostela
  - 659, Vigo
- Ukraine (7):
  - 791, Donetsk
  - 790, Kiev
  - 794, Kiev
  - 797, Kiev
  - 792, Luhansk
  - 793, Odesa
  - 796, Vinnytsia
- United Kingdom (3):
  - 677, Birmingham
  - 678, Christchurch
  - 679, London

REFERENCES:
- [Derived] Gottenberg JE, Dorner T, Bootsma H, Devauchelle-Pensec V, Bowman SJ, Mariette X, Bartz H, Oortgiesen M, Shock A, Koetse W, Galateanu C, Bongardt S, Wegener WA, Goldenberg DM, Meno-Tetang G, Kosutic G, Gordon C. Efficacy of Epratuzumab, an Anti-CD22 Monoclonal IgG Antibody, in Systemic Lupus Erythematosus Patients With Associated Sjogren's Syndrome: Post Hoc Analyses From the EMBODY Trials. Arthritis Rheumatol. 2018 May;70(5):763-773. doi: 10.1002/art.40425. Epub 2018 Apr 12. PMID 29381843
- [Derived] Clowse ME, Wallace DJ, Furie RA, Petri MA, Pike MC, Leszczynski P, Neuwelt CM, Hobbs K, Keiserman M, Duca L, Kalunian KC, Galateanu C, Bongardt S, Stach C, Beaudot C, Kilgallen B, Gordon C; EMBODY Investigator Group. Efficacy and Safety of Epratuzumab in Moderately to Severely Active Systemic Lupus Erythematosus: Results From Two Phase III Randomized, Double-Blind, Placebo-Controlled Trials. Arthritis Rheumatol. 2017 Feb;69(2):362-375. doi: 10.1002/art.39856. PMID 27598855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in December 2010 and concluded in June 2015.
Pre-assignment Details: Participant Flow refers to the Randomized Set (RS).
Groups:
- Placebo Weekly (RS): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 1200 mg Every Other Week (RS): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 600 mg Weekly (RS): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12 week treatment cycles
Period: Overall Study
Arm/Group | Placebo Weekly (RS) | Epratuzumab 1200 mg Every Other Week (RS) | Epratuzumab 600 mg Weekly (RS)
Started | 263 | 262 | 266
Completed | 178 | 171 | 184
Not Completed | 85 | 91 | 82
Not completed — Lack of Efficacy | 44 | 37 | 32
Not completed — Protocol Violation | 3 | 5 | 6
Not completed — Lost to Follow-up | 10 | 3 | 7
Not completed — Withdrawal by Subject | 12 | 14 | 14
Not completed — Death | 3 | 1 | 0
Not completed — Adverse Event | 9 | 24 | 19
Not completed — Patient non-availability | 1 | 1 | 1
Not completed — Suspected pregnancy | 1 | 1 | 0
Not completed — Patient non-compliance | 1 | 0 | 1
Not completed — Patient pregnant | 1 | 0 | 0
Not completed — Outside the study area | 0 | 2 | 1
Not completed — Lack of efficacy & patient not available | 0 | 1 | 0
Not completed — Patient withdrew after cardiology visit | 0 | 1 | 0
Not completed — Randomization error | 0 | 1 | 0
Not completed — Patient unable to start IV line | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to the Safety Set (SS).
Groups:
- Placebo Weekly (SS): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 1200 mg Every Other Week (SS): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 600 mg Weekly (SS): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12 week treatment cycles
Arm/Group | Placebo Weekly (SS) | Epratuzumab 1200 mg Every Other Week (SS) | Epratuzumab 600 mg Weekly (SS) | Total Title
Number analyzed (Participants) | 263 | 261 | 264 | 788
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 254 | 257 | 254 | 765
  >=65 years | 9 | 4 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (11.8) | 40.8 (11.5) | 41.2 (12.7) | 41.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 247 | 245 | 737
  Male | 18 | 14 | 19 | 51

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 48 According to a Combined Response Index
Description: Percentages are based on the number of subjects in the relevant treatment group within the Full Analysis Set (FAS). The combined response index incorporated criteria for achievement of responder status from the: British Isles Lupus Assessment Group Index (BILAG-2004)- improvement from study entry or no worsening in other organ systems, Systemic Lupus Erythematosus Disease Activity Index (SLEDAI; Version 2000, also known as SLEDAI-2K) - no worsening compared to study entry, physician's global assessment of disease activity(PGA)- no worsening compared to study entry, and concomitant medications- no changes.
Time Frame: At Week 48
Population: The Full Analysis Set (FAS) consisted of all subjects in the Randomized Set (RS) who had received at least 1 partial dose of the study drug.
Measure: Number; unit: Percentage of responders
Groups:
- Placebo Weekly (FAS): Placebo infusions delivered weekly for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 1200 mg Every Other Week (FAS): 1200 mg infusions delivered every other week for a total of 4 weeks (cumulative dose 2400 mg) over four 12-week treatment cycles and placebo infusions delivered every other week for a total of 4 weeks over four 12-week treatment cycles
- Epratuzumab 600 mg Weekly (FAS): 600 mg infusions delivered weekly for a total of 4 weeks (cumulative dose 2400 mg) over four 12 week treatment cycles
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of responders | 33.5 | 34.1 | 35.2
Statistical Analysis 1: Comparison: Placebo Weekly (FAS) vs Epratuzumab 1200 mg Every Other Week (FAS); Test type: Superiority; p = 0.899, Regression, Logistic — p-values for the comparison of treatment groups have been calculated using logistic regression with factors for treatment, pooled region, and baseline disease status; Odds Ratio (OR) = 1.024, 95% CI 2-sided [0.710 to 1.477] — Odds ratio: Epratuzumab/Placebo calculated using logistic regression with factors for treatment, pooled region, and baseline disease status
Statistical Analysis 2: Comparison: Placebo Weekly (FAS) vs Epratuzumab 600 mg Weekly (FAS); Test type: Superiority; p = 0.716, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.070, 95% CI 2-sided [0.743 to 1.539] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 24 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of responders | 32.3 | 33.0 | 43.6

3. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 12 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of responders | 30.0 | 32.2 | 40.9

4. Secondary Outcome: The Percent of Subjects Meeting Treatment Response Criteria at Week 36 According to a Combined Response Index
Description: as for outcome 1
Time Frame: At Week 36
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of responders | 32.7 | 33.0 | 36.7

5. Secondary Outcome: Change From Baseline in Daily Corticosteroid Dose at Week 24
Description: Participants were grouped into 4 categories: Dose decreased by >50%, Dose decreased >0% to ≤50%, No change in dose and Dose increased or missing data.
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of subjects
  Dose decreased by >50% | 4.6 (0) | 10.0 (0) | 8.7 (0)
  Dose decreased >0% to ≤50% | 20.9 (0) | 18.0 (0) | 18.2 (0)
  No change in dose | 48.3 (0) | 46.7 (0) | 52.7 (0)
  Dose increased or missing data | 26.2 (0) | 25.3 (0) | 20.5 (0)

6. Secondary Outcome: Change From Baseline in Daily Corticosteroid Dose at Week 48
Description: as for outcome 5
Time Frame: At Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Weekly (FAS) | Epratuzumab 1200 mg Every Other Week (FAS) | Epratuzumab 600 mg Weekly (FAS)
Number analyzed (Participants) | 263 | 261 | 264
Percentage of participants
  Dose decreased by >50% | 6.5 (0) | 13.8 (0) | 14.8 (0)
  Dose decreased >0% to ≤50% | 20.9 (0) | 13.4 (0) | 15.9 (0)
  No change in dose | 35.7 (0) | 35.6 (0) | 36.7 (0)
  Dose increased or missing data | 36.9 (0) | 37.2 (0) | 32.6 (0)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected throughout the study (on or after first infusion of study drug and within 75 days of the last infusion), for an average of 4.5 years (starting in December 2010 and concluding in June 2015). The Safety Set will be utilized for TEAE reporting.
Description: The Safety Set (SS) consisted of all subjects in the Randomized Set (RS) who had received at least 1 partial dose of study drug.
Arm/Group | Placebo Weekly (SS) | Epratuzumab 1200 mg Every Other Week (SS) | Epratuzumab 600 mg Weekly (SS)
All-Cause Mortality (participants affected / at risk) | 3/263 | 1/261 | 0/264
Serious Adverse Events (participants affected / at risk) | 45/263 | 45/261 | 50/264
Other Adverse Events (participants affected / at risk) | 151/263 | 145/261 | 158/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Weekly (SS) (N=263) | Epratuzumab 1200 mg Every Other Week (SS) (N=261) | Epratuzumab 600 mg Weekly (SS) (N=264)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lupus myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Necrotising retinitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 4 (5) | 3 (4)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection toxoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 6 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Lupus encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Noninfectious myelitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Weekly (SS) (N=263) | Epratuzumab 1200 mg Every Other Week (SS) (N=261) | Epratuzumab 600 mg Weekly (SS) (N=264)
Nausea (Gastrointestinal disorders) | 36 (51) | 32 (41) | 25 (38)
Diarrhoea (Gastrointestinal disorders) | 19 (24) | 15 (15) | 25 (41)
Vomiting (Gastrointestinal disorders) | 16 (18) | 12 (14) | 16 (23)
Fatigue (General disorders) | 14 (17) | 15 (31) | 15 (18)
Pyrexia (General disorders) | 17 (19) | 8 (9) | 13 (18)
Upper respiratory tract infection (Infections and infestations) | 37 (46) | 38 (49) | 37 (47)
Urinary tract infection (Infections and infestations) | 44 (66) | 37 (45) | 38 (54)
Nasopharyngitis (Infections and infestations) | 21 (23) | 15 (23) | 24 (31)
Sinusitis (Infections and infestations) | 19 (23) | 12 (17) | 20 (23)
Bronchitis (Infections and infestations) | 23 (24) | 13 (13) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (20) | 14 (16) | 14 (14)
Headache (Nervous system disorders) | 42 (68) | 29 (39) | 33 (50)
Dizziness (Nervous system disorders) | 13 (20) | 10 (15) | 14 (16)
Depression (Psychiatric disorders) | 15 (16) | 10 (11) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12) | 16 (19)
Hypertension (Vascular disorders) | 12 (12) | 13 (15) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days